CLINICAL TRIAL: NCT01504360
Title: Predictive Study of Radiation Induced Sarcoma From the GSF-GETO Data Base.
Brief Title: Predictive Study of Radiation Induced Sarcoma
Acronym: SARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0328-3maph11
Record Dates: First submitted 2011-12-30; First posted 2012-01-05 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2016-04

CONDITIONS: Radiation Induced Sarcoma
Keywords: sarcoma; radiation therapy; predictive essay
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sarcoma group (Experimental): patient suffering form radiation-induced sarcoma
  Interventions: Genetic: tumor genetic predisposition to develop sarcoma assessment
- free from sarcoma group (Active Comparator): patient without sarcoma 5 years after radiation therapy
  Interventions: Genetic: tumor genetic predisposition to develop sarcoma assessment

INTERVENTIONS:
Genetic: tumor genetic predisposition to develop sarcoma assessment — data concerning initial radiation and localisation of the sarcoma secondary developed will be collected. 2 blood samples (2 x 5 ml)will be collected. One sample of 5 mm will be dedicated to study radiation induced apoptosis assessed by flow cytometry. The second sample will be used to study the polymorphism of the genes involved in reparation of DNA by using chip screening of single nucleotide polymorphisms (SNP). DNA will be extracted and controlled by flow cytometrical separation.
  Arms: sarcoma group
Genetic: tumor genetic predisposition to develop sarcoma assessment — data concerning initial radiation and data demonstrating the lack of secondary sarcoma will be collected . 2 blood samples (2 x 5 ml)will be collected. One sample of 5 mm will be dedicated to study radiation induced apoptosis assessed by flow cytometry. The second sample will be used to study the polymorphism of the genes involved in reparation of DNA by using chip screening of single nucleotide polymorphisms (SNP). DNA will be extracted and controlled by flow cytometrical separation.
  Arms: free from sarcoma group

SUMMARY:
Development of sarcoma within or adjacent to radiation field is a well known event of poor prognosis and unknown risk factors. Advanced techniques of radiation therapy including intensity modulated radiation therapy, tomotherapy or Arc therapy are providing new modalities of radiation delivery that could be responsible for developing these induced tumors. There is little data on molecular biology of radiation induced sarcoma even if some tools are still available to characterize these types of tumors aiming to compare their profile to a sarcoma observed in non irradiated area. An update of the GETO-GCSF registry, currently called CONTICANET data base in the framework of EORTC, represents the backbone of the project. The next step should follow two axes, a clinical one based on the dosimetric analysis of the characteristics of delivered radiation therapy and the second one based on a molecular characterization of the sarcomas developed in irradiated field.The data base will be updated and organized through the CONTICANET network and the radiation oncologists involved in the treatment of soft tissue sarcoma. A retrospective analysis of the clinical data and the parameters describing the initial treatment will be registered using the methodology proposed by I. Diallo for radiation induced tumors developed in childhood. The most recent data will be extracted in DICOM format for intercomparison in a dedicated software.A centralized review of pathological specimens is planned to validate the correct classification of the tumors inside the current staging system developed for soft tissue sarcoma.

DETAILED DESCRIPTION:
The biological study will include the two following steps:1. On frozen specimen: genic profile of the tumor will be studied with two different techniques: CGH-array from extracted DNA in order to evaluate the number of gene copies, amplifications and deletions. The RNAm expression profile will be studied to evaluate the level of the gene expression. More than 200 data collected in Institut Bergonié, coming from de novo sarcoma would be used as a comparative specimen since the pathological diagnosis is the same as the one observed for radiation induced sarcoma. A comparison between the two populations will be able to define profiles, gene modifications and signalisation pathways of radiation induced sarcoma. 2. On blood sample: 2 groups of patients will be compared: those with radiation induced sarcoma and patients receiving radiation therapy for more than 5 years ago without developing sarcoma. The study will be performed with the inform consent of the patients and of the controlled cases.This second step requires 2 blood samples (2 x 5 ml). They will be collected and sent to the molecular biology laboratory located in Centre Alexis VAUTRIN (Nancy).- One sample of 5 mm will be dedicated to study radiation induced apoptosis assessed by flow cytometry. A correlation has been described between radiation-induced apoptosis of CT8+ lymphocytes after an 8 Gy irradiation and the occurrence of severe late toxicity after radiation therapy for patients treated for several types of tumors.- The second sample will be used to study the polymorphism of the genes involved in reparation of DNA by using chip screening of single nucleotide polymorphisms (SNP). This sample will be used after DNA extraction from mononuclear blood cells. DNA will be extracted and controlled by flow cytometrical separation. It will be sent to Bordeaux molecular biology laboratory in Institut Bergonié (Prof. JM COINDRE) to perform an evaluation of the single nucleotide polymorphism. The aim of this part of the protocol is to study variances in gene, the product of which plays a role in radiation response and in the development of adverse effects after radiation therapy. For patients with radiation-induced sarcoma, the results of this analysis will be compared with the data obtained from DNA analysis extracted from the tumors. The clinical, pathological and biological characterisation of radiation-induced sarcoma obtained will allow to identify constitutional variances linked with an increased sensitivity to radiation therapy leading to discuss indication of irradiation in a population at risk. Pediatric radiation therapy and adjuvant treatment after surgery for breast carcinoma will be the main targets of this selection of patients. This project will be able to select radiation modality in patients at risk (intensity modulated radiation therapy or 3D conformal approach, stereotactic approaches, partial irradiation of the breast).

ELIGIBILITY:
radiation-induced sarcoma group

Inclusion Criteria:

1. Age > 18 ans when radiation was performed
2. suffering from a radiation induced sarcoma

Exclusion Criteria:

1. private individuals of freedom or under tutelage (including legal guardianship)
2. initial tumor treated by radiotherapy was a sarcoma
3. patient bearer of an osteosarcoma

Free from irradiation induced sarcoma group

Inclusion Criteria:

1. Age > 18 ans when radiation was performed
2. surviving irradiated patients for cancer for more than 5 years and free of from radiation-induced sarcoma.

Exclusion Criteria:

1. private individuals of freedom or under tutelage (including legal guardianship)
2. History of cancer (except baso-cellular cutaneous epithelioma or in situ epithelioma of the cervix) that has relapsed in the 5 years preceding recruitment for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2011-12; Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Determine the predictive clinical and biological risk factors to develop a sarcoma on irradiated territory. | from date of inclusion up to the end of recruiting period : november 2013 (anticipated)
  Clinical data of initial radiation therapy, radiation-induced apoptosis of CT8+ lymphocytes and polymorphism of the genes involved in reparation of DNA by using chip screening of single nucleotide polymorphisms (SNP) will be studied for each patient included.

CONTACTS AND LOCATIONS:
Overall Officials: Phillipe Maingon, Professor, Principal Investigator — Centre Georges Francois Leclerc
Locations (1):
- CGFL, Dijon, France